CLINICAL TRIAL: NCT00876915
Title: A Prospective Randomized Multicenter Study of Dalteparin Prophylaxis in High-Risk Ambulatory Cancer Patients
Brief Title: A Study of Dalteparin Prophylaxis in High-Risk Ambulatory Cancer Patients
Acronym: PHACS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow enrollment and lack of continuing funds
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Charles Francis, Professor emeritus, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25387; 1R01HL095109-01 (NIH)
Record Dates: First submitted 2009-03-31; First posted 2009-04-07 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism
Keywords: prevention of VTE and PE in high risk cancer patients
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Risk for VTE recieving dalteparin (Experimental): Patients assigned at random to receive prophylactic dalteparin injections
  Interventions: Drug: dalteparin injection
- High Risk for VTE No therapy (No Intervention): No prophylactic therapy for VTE prevention given (Subjects receiving standard of care)
- Low Risk for VTE (No Intervention): Used as a control for the secondary outcome of evaluating tissue factor in collected blood samples

INTERVENTIONS:
Drug: dalteparin injection — Potency is described in international anti-Xa units (IU). One unit (anti-Xa) of dalteparin sodium, average molecular weight 5,000, corresponds to the activity of one unit of the 1st International Standard for Low Molecular Weight Heparin (LMWH)with respect to inhibition of coagulation Factor Xa in plasma utilizing the chromogenic peptide substrate S-2765 (N-alpha-Benzyloxycarbonyl-D-arginyl-glycyl-arginine-pNA.2HCl).
  Other Names: Fragmin
  Arms: High Risk for VTE recieving dalteparin

SUMMARY:
Some cancer patients starting a new chemotherapy regimen are likely to develop blood clots, also known as venous thromboembolism (VTE). Blood clots can cause symptoms and can occasionally be life-threatening. The purpose of this study is to determine if a daily injection of a blood-thinner, dalteparin, for 12 weeks can safely and effectively reduce the frequency of blood clots. Dalteparin is currently approved for prevention of blood clots following surgery and in hospitalized patients but not specifically for cancer outpatients.

DETAILED DESCRIPTION:
VTE is an increasingly frequent complication of cancer and anti-cancer therapies. It is associated with increased mortality and other significant adverse consequences. Risk factors for VTE in the cancer population have been identified, and multiple studies have also shown that VTE can be prevented in high-risk populations with the use of thromboprophylaxis. This study evaluated the safety and efficacy of prophylaxis in a high-risk subgroup of cancer patients identified by a validated risk model developed by us previously called the "Khorana Score." Correlative studies evaluated the value of tissue factor as a predictive biomarker of VTE. The purpose of this study was to conduct a prospective, randomized clinical trial comparing the safety and efficacy of prophylaxis with dalteparin to no treatment in reducing VTE in high-risk ambulatory cancer patients initiating chemotherapy and to establish the value of TF as a predictive marker for VTE in ambulatory cancer patients receiving chemotherapy.

PHACS was a randomized multi-center clinical trial. Eligible patients were enrolled and underwent baseline screening ultrasonography of the lower extremities to rule out pre-existing DVT and a chest CT scan to rule out PE. If negative, patients were then randomized to receive either dalteparin 5000 units subcutaneously daily or observation for a study period of 12 weeks. The first day of dalteparin prophylaxis coincided with the first day of initiation of a new systemic chemotherapy regimen. The patients were seen every 4 weeks (±1 week) at the time of regularly scheduled chemotherapy cycle visits for serial ultrasonography of lower extremities during study period (i.e. at 4, 8 and 12 weeks.) A chest CT scan was performed at 12 weeks. Compliance was measured by asking patients about missed doses at these 4-weekly visits as well as by asking patients to fill an injection diary.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of malignancy;
* At planned initiation of a new systemic chemotherapy regimen (including patients starting on first chemotherapy or patients previously treated but starting on a new regimen);
* A risk score for VTE ≥3 [assign score of 2 for very high risk sites of cancer (stomach, pancreas), score of 1 for high risk site (lung, lymphoma, gynecologic, bladder, testicular) and score of 0 for all other sites], hemoglobin <10 g/dL or planned use of erythropoiesis stimulating agents, platelet count ≥350,000/mm3, total leukocyte count > 11,000/mm3 or body mass index ≥ 35 kg/m2]. Any counts meeting criteria drawn within 2 weeks prior to enrollment are considered acceptable.
* Age 18 years or older
* Provide written, informed consent.

Exclusion Criteria:

* Active bleeding or at high risk of serious bleeding complication in the opinion of the investigator
* Diagnosis of primary brain tumor multiple myeloma, leukemia, or myelodysplastic syndrome
* Planned stem cell transplant
* Life expectancy < 6 months
* Known allergy to heparin or LMWH
* Patient or caregiver incapable of daily self-injection
* Acute or chronic renal insufficiency with creatinine clearance < 30 mL/min
* History of heparin-induced thrombocytopenia
* Allergy to contrast agents
* Pregnancy
* Need for anticoagulant therapy
* Platelet count < 75,000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W. Francis, MD, Principal Investigator — Univeristy of Rochester Medical Center
Locations (7):
- United States (6):
  - University of California, Davis, Sacramento, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- Ottawa Hospital Research Institute (OHRI), Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Khorana AA, Francis CW, Kuderer NM, Carrier M, Ortel TL, Wun T, Rubens D, Hobbs S, Iyer R, Peterson D, Baran A, Kaproth-Joslin K, Lyman GH. Dalteparin thromboprophylaxis in cancer patients at high risk for venous thromboembolism: A randomized trial. Thromb Res. 2017 Mar;151:89-95. doi: 10.1016/j.thromres.2017.01.009. Epub 2017 Jan 26. PMID 28139259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants screened for the study but deemed low or medium risk by Khorona scoring will be offered to consent to a one time baseline blood sample. These samples will be used as the control group to establish the value of TF as a predictive marker for VTE in ambulatory cancer patients as described in the Secondary Objectives.
Pre-assignment Details: Participants who undergo a baseline US/CT scan and are found to have a DVT/PE will be considered a screen failure and will not be randomized and continue on in the study. In addition, if any of the screening criteria are not met, these subjects will be considered screen failures.
Groups:
- High Risk Dalteparin Injection: Patients will be assigned at random to receive prophylactic dalteparin injections
  dalteparin injection: Potency is described in international anti-Xa units (IU). One unit (anti-Xa) of dalteparin sodium, average molecular weight 5,000, corresponds to the activity of one unit of the 1st International Standard for Low Molecular Weight Heparin (LMWH)with respect to inhibition of coagulation Factor Xa in plasma utilizing the chromogenic peptide substrate S-2765 (N-alpha-Benzyloxycarbonyl-D-arginyl-glycyl-arginine-pNA.2HCl).
- High Risk No Therapy: No prophylactic therapy for VTE prevention given (Subjects just receiving standard of care)
- Low or Medium Risk Group: Subjects deemed low or medium risk for VTE by Khorona score. These subjects did not enter into the study but supplied a one-time baseline blood sample for use as a control in the studies Secondary Objective of establishing the value of TF as a predictive marker for VTE.
Period: Overall Study
Arm/Group | High Risk Dalteparin Injection | High Risk No Therapy | Low or Medium Risk Group
Started | 50 | 48 | 101
Week 4 | 38 | 45 | 0
Week 8 | 33 | 36 | 0
Completed | 31 | 34 | 101
Not Completed | 19 | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Risk Randomized to Dalteparin Injection: Patients will be assigned at random to receive prophylactic dalteparin injections
  dalteparin injection: Potency is described in international anti-Xa units (IU). One unit (anti-Xa) of dalteparin sodium, average molecular weight 5,000, corresponds to the activity of one unit of the 1st International Standard for Low Molecular Weight Heparin (LMWH)with respect to inhibition of coagulation Factor Xa in plasma utilizing the chromogenic peptide substrate S-2765 (N-alpha-Benzyloxycarbonyl-D-arginyl-glycyl-arginine-pNA.2HCl).
- High Risk Randomized to No Therapy: No prophylactic therapy for VTE prevention given (Subjects just receiving standard of care)
- Low Risk: Ambulatory cancer patients deemed Low risk based on a Khorona score of 0-2
- Total: Total of all reporting groups
Arm/Group | High Risk Randomized to Dalteparin Injection | High Risk Randomized to No Therapy | Low Risk | Total
Number analyzed (Participants) | 50 | 48 | 101 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 35 | 74 | 143
  >=65 years | 16 | 13 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 58 (12) | 58 (13) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 41 | 86
  Male | 29 | 24 | 60 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 48 | 45 | 96 | 189
  Unknown or Not Reported | 0 | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 4
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 7 | 8 | 9 | 24
  White | 38 | 37 | 91 | 166
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 0 | 7
  United States | 46 | 45 | 101 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Venous Thromboembolisms
Description: The percentage of patients who developed a Venous thromboembolism were recorded within 12 weeks following randomization including all adjudicated occurrences of symptomatic DVT, PE and upper extremity thrombus as well as all asymptomatic DVT and PE detected by lower extremity ultrasonography and chest CT.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Groups:
- Dalteparin Injection: Patients will be assigned at random to receive prophylactic dalteparin injections
  dalteparin injection: Potency is described in international anti-Xa units (IU). One unit (anti-Xa) of dalteparin sodium, average molecular weight 5,000, corresponds to the activity of one unit of the 1st International Standard for Low Molecular Weight Heparin (LMWH)with respect to inhibition of coagulation Factor Xa in plasma utilizing the chromogenic peptide substrate S-2765 (N-alpha-Benzyloxycarbonyl-D-arginyl-glycyl-arginine-pNA.2HCl).
- No Therapy: No prophylactic therapy for VTE prevention given (Subjects just receiving standard of care)
Arm/Group | Dalteparin Injection | No Therapy
Number analyzed (Participants) | 50 | 48
percentage of participants | 12 | 21
Statistical Analysis 1: Comparison: Dalteparin Injection vs No Therapy; Test type: Superiority or Other; p = 0.4795, stratified Cox; Hazard Ratio (HR) = 0.695, 95% CI 2-sided [0.235 to 1.890]

2. Primary Outcome: Percentage of Patients Who Experienced Clinically Significant Bleeding Events.
Description: The percentage of patients who experienced a clinically significant bleeding event were recorded (including major and clinically significant non-major bleeding) over 13 weeks (12 weeks of study and an additional week of observation). Major bleeding was defined as being clinically overt and satisfying one of the following: decrease in hemoglobin of 2.0 g/dL, leading to transfusion of 2 or more units of blood or packed red cells, occurring in a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial) or leading to death. Clinically significant non-major bleeding was defined as clinically overt, not meeting criteria for major bleeding and with one of the following characteristics: multiple-source, spontaneous hematoma > 25 cm², epistaxis > 5 mins, macroscopic hematuria not related to instrumentation, spontaneous rectal bleeding, gingival bleeding > 5 mins, hemoptysis, hematemesis or prolonged bleeding (> 5 minutes) after venipuncture.
Time Frame: 13 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Dalteparin Injection | No Therapy
Number analyzed (Participants) | 50 | 48
percentage of participants | 14 | 2
Statistical Analysis 1: Comparison: Dalteparin Injection vs No Therapy; Test type: Superiority or Other; p = 0.0252, stratified Cox; Hazard Ratio (HR) = 7.019, 95% CI 2-sided [1.236 to 131.632]

3. Secondary Outcome: The Value of Tissue Factor (TF) at Baseline Prior to Chemotherapy in Ambulatory Cancer Patients
Description: Blood samples were obtained to measure the value of Tissue Factor at baseline compared between high risk for VTE and low risk for VTE ambulatory cancer patients.
Time Frame: baseline value of tissue factor
Population: From 98 high risk patients, 89 provided blood samples used for this analysis. From the low risk group, all 101 subjects provided blood samples for analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- High Risk: High Risk participants ambulatory cancer patients with Khorona scores 3+
- Low Risk: Low Risk ambulatory cancer patients with Khorona scores of 0-2
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 89 | 101
pg/mL | 0.669 (1.35) | 0.187 (0.492)

4. Secondary Outcome: The Value of D-Dimer at Baseline Prior to Chemotherapy in Ambulatory Cancer Patients
Description: Blood samples were obtained to measure the value of D-Dimer at baseline compared between high risk for VTE and low risk for VTE ambulatory cancer patients
Time Frame: baseline value of D-Dimer
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 89 | 101
ug/mL | 2.99 (5.67) | 1.87 (3.67)

5. Secondary Outcome: The Value of Human F12 at Baseline Prior to Chemotherapy in Ambulatory Cancer Patients
Description: Blood samples were obtained to measure the value of Human F12 at baseline compared between high risk for VTE and low risk for VTE ambulatory cancer patients
Time Frame: baseline value of Human F12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 89 | 101
ng/mL | 484.7 (1167.6) | 306.3 (552.7)

6. Secondary Outcome: The Value of Tissue Factor Pathway Inhibitor (TFPI) at Baseline Prior to Chemotherapy in Ambulatory Cancer Patients
Description: Blood samples were obtained to measure the value of TFPI at baseline compared between high risk for VTE and low risk for VTE ambulatory cancer patients
Time Frame: baseline value of TFPI
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 89 | 101
pg/mL | 813.6 (391.3) | 738.2 (351.1)

7. Secondary Outcome: The Value of Factor VIIa (FVIIa) at Baseline Prior to Chemotherapy in Ambulatory Cancer Patients
Description: Blood samples were obtained to measure the value of FVIIa at baseline compared between high risk for VTE and low risk for VTE ambulatory cancer patients
Time Frame: baseline value of FVIIa
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pM
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 89 | 101
pM | 151.2 (59.4) | 148.6 (92.2)

8. Secondary Outcome: The Value of Thrombin Antithrombin (TAT) at Baseline Prior to Chemotherapy in Ambulatory Cancer Patients
Description: Blood samples were obtained to measure the value of TAT at baseline compared between high risk for VTE and low risk for VTE ambulatory cancer patients
Time Frame: baseline value of TAT
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | High Risk | Low Risk
Number analyzed (Participants) | 89 | 101
ug/L | 9.89 (20.09) | 12.44 (21.42)

ADVERSE EVENTS:
Time Frame: 13 weeks, 12 weeks on active treatment + 1 additional week
Arm/Group | Dalteparin Injection | No Therapy
Serious Adverse Events (participants affected / at risk) | 26/50 | 18/48
Other Adverse Events (participants affected / at risk) | 39/50 | 43/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalteparin Injection (N=50) | No Therapy (N=48)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiac Troponin T (Cardiac disorders) | 1 (1) | 0 (0)
bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cholangitis-bilary tree stricture (Gastrointestinal disorders) | 0 (0) | 2 (2)
Confusion (Social circumstances) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Death (Investigations) | 2 (2) | 1 (1)
Dehydration (Gastrointestinal disorders) | 4 (5) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 3 (3) | 1 (1)
febrile neutropenia (Infections and infestations) | 3 (3) | 1 (1)
Fever (General disorders) | 1 (1) | 3 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Obstruction - biliary tree (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Glucose, serum - high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose, serum - low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 (0) | 2 (6)
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 4 (4) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Infection - Other (Sepsis) (Infections and infestations) | 2 (2) | 3 (3)
Infection - Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (Spontaneous Bacterial Peritonitis) (Infections and infestations) | 0 (0) | 1 (1)
Infection - Other (Infections and infestations) | 2 (2) | 0 (0)
Infection - Other (skin cellulitis) (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC (Infections and infestations) | 3 (3) | 2 (2)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Mucositis (functional/symptomatic) - oral cavity (Gastrointestinal disorders) | 1 (1) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness - whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (2)
Neurology - Other (altered mental status) (Psychiatric disorders) | 0 (0) | 2 (2)
Neurology - Other (loss of consciousness) (Nervous system disorders) | 0 (0) | 1 (1)
Neurology - Other (pseudoseizures) (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy - motor (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Abdomen NOS (Gastrointestinal disorders) | 4 (5) | 3 (5)
Pain - chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pain - Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - head/headache (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - NOS (General disorders) | 1 (1) | 0 (0)
Perforation, GI (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Potassium, serum - high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
sodium, serum - low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Somnolence/depressed level of consciousness (Psychiatric disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 1 (1)
Thrombosis/Thrombus/embolism (Vascular disorders) | 3 (3) | 1 (1)
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (3)
Ventricular arrhythmia - ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalteparin Injection (N=50) | No Therapy (N=48)
Albumin, serum - low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (7) | 8 (8)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3 (3) | 8 (9)
allergic reaction/hypersensetivity (General disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ALT (Metabolism and nutrition disorders) | 13 (13) | 10 (11)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (9) | 12 (12)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
AST (Metabolism and nutrition disorders) | 9 (9) | 13 (16)
bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
blood - other (leukocytosis) (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
bruising (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
calcium, serum - high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
calcium, serum - low (hypocalcemia) (Metabolism and nutrition disorders) | 8 (8) | 8 (8)
confusion (Psychiatric disorders) | 3 (5) | 2 (2)
colitis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 13 (13) | 7 (8)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
constitutional symptoms - other (cachexia) (General disorders) | 0 (0) | 1 (1)
creatinine (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
diarrhea (Metabolism and nutrition disorders) | 9 (12) | 13 (15)
dizziness (Nervous system disorders) | 3 (3) | 8 (8)
distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1)
dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
edema: limb (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 18 (18) | 21 (24)
febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0)
fever (Infections and infestations) | 11 (12) | 3 (3)
flu-like symptoms (Infections and infestations) | 3 (3) | 1 (1)
flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
glucose, serum - high (hyperglycemia) (Metabolism and nutrition disorders) | 11 (11) | 10 (11)
glucose, serum - low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
gastrointestinal - incontinence, bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI - other (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI - other (biliary tree obstruction) (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastrointestinal - other (gas pain) (Gastrointestinal disorders) | 1 (1) | 0 (0)
heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
hemoglobin (Blood and lymphatic system disorders) | 17 (21) | 20 (21)
henorrhage, GI - Rectum (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemorrhage, pulmonary/upper respiratory - nose (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
hemorrhage, GI-Lower GI NOS (Gastrointestinal disorders) | 1 (2) | 0 (0)
hemorrhage, GI-upper GI NOS (Gastrointestinal disorders) | 1 (2) | 0 (0)
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 1 (1)
hypotension (Cardiac disorders) | 5 (6) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
infection - conjunctiva (Infections and infestations) | 0 (0) | 1 (1)
infection - other (sinus) (Infections and infestations) | 1 (1) | 0 (0)
infection - other (Infections and infestations) | 0 (0) | 1 (1)
infection - other (skin, cellulitis) (Infections and infestations) | 0 (0) | 1 (1)
infection - other (thrush) (Infections and infestations) | 2 (3) | 2 (2)
infection - other (urinary tract NOS) (Infections and infestations) | 1 (1) | 1 (1)
infection - other (upper respiratory) (Infections and infestations) | 1 (1) | 0 (0)
infection with grade 2 neutrophils - skin (cellulitis) (Infections and infestations) | 0 (0) | 1 (1)
infection with normal ANC (Infections and infestations) | 2 (2) | 0 (0)
infection with normal ANC - bronchus (Infections and infestations) | 1 (1) | 0 (0)
infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
insomnia (General disorders) | 4 (4) | 4 (4)
leukocytes (total WBC) (Blood and lymphatic system disorders) | 13 (13) | 14 (17)
liver dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
lymphatics - other (anasarca) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
magnesium, serum - low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
memory impairment (Psychiatric disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 20 (22) | 23 (25)
neuropathy - sensory (Nervous system disorders) | 2 (2) | 15 (15)
neurology - other (neuropraxia) (Nervous system disorders) | 1 (1) | 0 (0)
neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10 (10) | 10 (11)
obstruction - Gtube (Gastrointestinal disorders) | 0 (0) | 1 (1)
pain - abdomen NOS (General disorders) | 8 (9) | 7 (7)
platelets (Blood and lymphatic system disorders) | 7 (7) | 10 (11)
vomiting (Gastrointestinal disorders) | 7 (8) | 15 (17)
weight loss (General disorders) | 11 (11) | 10 (10)
potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (6) | 2 (4)
potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (3) | 6 (7)
pain - chest/thorax NOS (General disorders) | 1 (1) | 0 (0)
pain - back (General disorders) | 0 (0) | 1 (1)
pain - dysuria (painful urination) (Renal and urinary disorders) | 2 (2) | 0 (0)
pain - throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
pain - extremity - limb (General disorders) | 3 (3) | 2 (3)
pain - cardiac/chest (Cardiac disorders) | 0 (0) | 1 (1)
pain - head/headache (General disorders) | 3 (3) | 2 (2)
pain - muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
pain - other (ear) (Ear and labyrinth disorders) | 1 (1) | 1 (1)
pain - other (groin) (General disorders) | 0 (0) | 1 (1)
pain - joint (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
pain - other (jaw) (General disorders) | 0 (0) | 1 (1)
pain - NOS (General disorders) | 1 (1) | 0 (0)
pain - other (knee) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain - other (peg tube site) (General disorders) | 0 (0) | 1 (1)
pain - skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pain - stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
phlebitis (Vascular disorders) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
psychosis (hallucinations/delusions) (Psychiatric disorders) | 3 (3) | 1 (1)
rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
rigors/chills (General disorders) | 3 (3) | 4 (5)
salivary gland changes/saliva (Gastrointestinal disorders) | 1 (1) | 1 (1)
sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
skin breakdown (thighs) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
supraventricular arrythmia - sinus tachycardia (Cardiac disorders) | 3 (3) | 4 (4)
supraventricular arrythmia - atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
mood alteration - agitation (Psychiatric disorders) | 3 (3) | 0 (0)
metabolic/laboratory - other (azotemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
mood alteration - anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
mood alteration - depression (Psychiatric disorders) | 0 (0) | 1 (1)
mucositis (fuctional/symptomatic) - oral cavity (Gastrointestinal disorders) | 2 (2) | 4 (4)
dermatitis - chemoradiation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
muscle weakness - whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 2 (2)
syndromes - other (serotonergic syndrome) (Endocrine disorders) | 1 (1) | 0 (0)
syndromes - other (systemic inflammatory response syndrome (SIRS)) (Infections and infestations) | 1 (1) | 0 (0)
taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 3 (3)
tremor (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 6 (6)
ulcer, GI - stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
vascular - thrombosis (Vascular disorders) | 1 (1) | 2 (2)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 2 (2)
ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
voice changes (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No